CLINICAL TRIAL: NCT06937424
Title: Effectiveness of Post-Endodontic Access-Cavity Cleaning Techniques: A Randomized Clinical Study
Brief Title: Post-endodontic Access Cavity Cleaning Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/22/983
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Teeth With Root Canal Treatment
Keywords: sealer; contamination; cleaning; air polishing; air abrasion; microbrush
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- • Dry cotton pellet group (Experimental): The contaminated dentine surface was scrubbed with a dry cotton pellet until no visible sealer remnants were observed
  Interventions: Other: Dry cotton pellet group
- Ethanol-saturated cotton pellet 7 seconds group (Experimental): The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet for 7 seconds
  Interventions: Other: Ethanol-saturated cotton pellet 7 seconds group
- Ethanol-saturated cotton pellet visibly clean group (Experimental): The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed.
  Interventions: Other: Ethanol-saturated cotton pellet visibly clean group
- Ethanol-saturated cotton Pellet + air polishing group (Experimental): After the contaminated dentine surface scrubbing with an 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed, air polishing was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Sodium bicarbonate powder (Velopex) was applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.
  Interventions: Device: Ethanol-saturated cotton Pellet + air polishing group
- Microbrush 7 sec group (Experimental): The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush for 7 seconds
  Interventions: Other: Microbrush 7 sec group
- Microbrush visibly clean group (Experimental): The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush until no visible sealer remnants were observed.
  Interventions: Other: Microbrush visibly clean group
- Air abrasion group (Experimental): Air abrasion was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Aluminium oxide particles (53 µm, Velopex) were applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.
  Interventions: Device: Air abrasion group

INTERVENTIONS:
Other: Dry cotton pellet group — The contaminated dentine surface was scrubbed with a dry cotton pellet until no visible sealer remnants were observed
  Arms: • Dry cotton pellet group
Other: Ethanol-saturated cotton pellet 7 seconds group — The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet for 7 seconds
  Arms: Ethanol-saturated cotton pellet 7 seconds group
Other: Ethanol-saturated cotton pellet visibly clean group — The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed.
  Arms: Ethanol-saturated cotton pellet visibly clean group
Device: Ethanol-saturated cotton Pellet + air polishing group — After the contaminated dentine surface scrubbing with an 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed, air polishing was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Sodium bicarbonate powder (Velopex) was applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.
  Arms: Ethanol-saturated cotton Pellet + air polishing group
Other: Microbrush 7 sec group — The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush for 7 seconds
  Arms: Microbrush 7 sec group
Other: Microbrush visibly clean group — The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush until no visible sealer remnants were observed.
  Arms: Microbrush visibly clean group
Device: Air abrasion group — Air abrasion was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Aluminium oxide particles (53 µm, Velopex) were applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.
  Arms: Air abrasion group

SUMMARY:
Aim This study aims to evaluate the effectiveness of different post-endodontic access cavity cleaning techniques (PACCTs) in removing residual epoxy resin-based root canal sealer from the pulp chamber floor following root canal treatment. The cleaning efficacy of seven different protocols, including manual and mechanically-assisted methods, will be compared based on the reduction of sealer-covered area (SCA).

Study Design / Methodology This study is designed as a prospective, single-center, randomized clinical trial with parallel group design.

A total of 70 patients who require root canal treatment in maxillary first molars will be included in the study. Patients will be randomly assigned to seven experimental groups (n=10 per group) according to the cleaning technique used after root canal obturation with AH Plus epoxy resin-based sealer.

The cleaning protocols will be:

1. Dry cotton pellet (control group)
2. Ethanol-saturated cotton pellet (7 sec)
3. Ethanol-saturated cotton pellet (visibly clean)
4. Ethanol-saturated cotton pellet + air polishing
5. Ethanol-saturated microbrush (7 sec)
6. Ethanol-saturated microbrush (visibly clean)
7. Air abrasion Standard root canal treatment procedures will be performed in all groups using rotary instrumentation and cold lateral condensation technique for obturation.

The cleaning effectiveness will be evaluated using standardized high-resolution macro photographs taken before and after the cleaning procedures. The sealer-covered area (SCA) will be calculated using image analysis software (Adobe Photoshop) based on pixel analysis.

The primary outcome of the study is the percentage reduction of SCA after cleaning procedures.

DETAILED DESCRIPTION:
Study design The study protocol was approved by the Committee of Research Ethics under the protocol number 2024/22/983. This study has been registered with clinicaltrials.gov under the title: Effectiveness of Post-Endodontic Access-Cavity Cleaning Techniques (PACCTs): A Randomized Clinical Study with an identifier: ….. The present randomized clinical trial was conducted and reported in accordance with the 2020 PRIRATE (Preferred Reporting Items for Randomized Trials in Endodontics) guidelines (Nagendrababu et al., 2020). All clinical procedures were conducted in accordance with the principles of good clinical practice and the ethical standards outlined in the Declaration of Helsinki. The design of the study is presented in Figure 1.

Sample size Power analysis was performed using G*Power software (Version XX, University of Düsseldorf, Germany). In the absence of available clinical data in the literature, the sample size calculation was based on the findings of a pilot study. With an effect size of 0.8 and an alpha error probability of 0.05, the power of the study was estimated to exceed 80%, and the total sample size was determined as 35.

Inclusion and exclusion criteria Systemically healthy patients aged between 18 and 65 years who required routine root canal treatment in maxillary first molars were included in the study. Additional inclusion criteria were as follows: patients with sufficient cognitive ability to understand and provide informed consent, teeth undergoing primary root canal treatment, and cases in which the use of an AH Plus epoxy resin-based sealer was deemed appropriate. Exclusion criteria were as follows: teeth with a history of previous root canal treatment; patients with systemic diseases, known allergies, or pregnancy; patients who refused to participate or did not provide informed consent; teeth with unclear visualization of the cavity floor; and cases in which the access cavity design or cleaning protocol could not be standardized.

Randomization and allocation concealment Patients were randomly assigned to seven experimental groups using a computer-generated random sequence (www.randomizer.org). The allocation sequence was prepared by an independent researcher who was not involved in the treatment procedures. Group assignment was concealed in sealed opaque envelopes and revealed immediately before the intervention.

Root canal treatment protocol All root canal treatments were performed by a single endodontist with more than five years of clinical experience. Local anaesthesia was administered using 2% articaine with 1:100,000 epinephrine (Ultracaine D-S Forte, Hoechst Marion Roussel, Germany). Following rubber dam isolation, standard access cavities were prepared using high-speed diamond burs under water cooling. All procedures were carried out under dental magnification with 5.7× loupes (ExamVision, Denmark). Working length was determined using an electronic apex locator (Root ZX II, Morita, Tokyo, Japan) and confirmed radiographically. Root canal instrumentation was performed using a rotary NiTi system (FKG Dentaire, La Chaux-de-Fonds, Switzerland) in accordance with the manufacturer's instructions. Irrigation was performed using 2.5% sodium hypochlorite (NaOCl) throughout the instrumentation. Final irrigation was performed using 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) for 1 minute, followed by a final flush with 5 mL of distilled water. Ultrasonic activation of the irrigants was applied during the final irrigation phase using an ultrasonic unit (Piezon Master 700, EMS, Nyon, Switzerland) to enhance the removal of debris and smear layer. After drying the canals with sterile paper points, root canal obturation was performed using the cold lateral condensation technique with gutta-percha cones and an epoxy resin-based sealer (AH Plus, Dentsply DeTrey, Konstanz, Germany). The sealer was applied to the canal walls using the master cone. Following obturation, the excess gutta-percha was removed with a heated instrument at the canal orifice level, and vertical compaction was applied. All treatments were performed following a standardized protocol to minimize operator-dependent variability and ensure consistency across all cases.

Cleaning Protocol Seven different cleaning methods were performed to remove the sealer-contaminated dentine.

* Dry cotton pellet group: The contaminated dentine surface was scrubbed with a dry cotton pellet until no visible sealer remnants were observed (previous studies: Ulusoy et al. 2016; da Silva et al. 2020).
* Ethanol-saturated cotton pellet 7 seconds group: The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet for 7 seconds (Ulusoy et al. 2016; da Silva et al. 2020).
* Ethanol-saturated cotton pellet visibly clean group: The contaminated dentine surface was scrubbed with a 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed.
* Ethanol-saturated cotton Pellet + air polishing group: After the contaminated dentine surface scrubbing with an 70% ethanol-saturated cotton pellet until no visible sealer remnants were observed, air polishing was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Sodium bicarbonate powder (Velopex) was applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.
* Microbrush 7 sec group: The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush for 7 seconds (Ulusoy et al. 2016).
* Microbrush visibly clean group: The contaminated dentine surface was scrubbed with a 70% ethanol-saturated microbrush until no visible sealer remnants were observed.
* Air abrasion group: Air abrasion was performed for 10 seconds using the AquaCare Twin device (Velopex, UK). Aluminium oxide particles (53 µm, Velopex) were applied at a pressure of 2 bar, with a medium media flow and 17.5% ethanol-saturated solution (AquaSol, Velopex). The standard tip was positioned approximately 5 mm from the dentin surface and moved in a vertical (up-and-down) direction during the procedure. The application time and parameters were determined in consultation with the manufacturer due to the lack of previous clinical studies using the AquaCare device for this purpose.

Following all cleaning procedures, an air/water spray was applied to the cavity surface to remove any remaining particles or cleaning agents.

Assessment Protocol The cleaning effectiveness at the cavity floor was assessed using standardized macro photographs of the cavity surfaces. Standardized photographs were taken immediately after the root canal obturation (pre-cleaning) and repeated following the completion of the cleaning procedures (post-cleaning). All images were captured using a digital single-lens reflex (DSLR) camera (Nikon D750, Nikon Corporation, Tokyo, Japan) equipped with a 105 mm macro lens (AF-S VR Micro-Nikkor 105 mm f/2.8G IF-ED, Nikon Corporation, Tokyo, Japan) and a paraflash lighting system (Visico, China) to ensure optimal standardization and illumination conditions. The shooting parameters were set at shutter speed 1/125, aperture f/2.8, ISO 200.

The measurements were performed by a single experienced researcher who was blinded to the cleaning protocols applied to the specimens. The photographs were quantitatively analyzed using image analysis software (Photoshop CC, Adobe Systems Inc., San Jose, CA, USA).

In the software, the cavity floor surface areas were selected using the quick selection tool, and the number of pixels corresponding to the residual sealer was calculated. The number of pixels within the encircled area was determined using the histogram tool. The ratio of the sealer-contaminated area to the total cavity floor area was determined and recorded as a percentage for each specimen (Figure X). To ensure measurement reliability, the assessment was repeated three times for each image, and all measurements were recorded.

Statistical analysis Statistical analysis was performed using SPSS software (Version XX, IBM Corp., Armonk, NY, USA). Initially, the normality of data distribution was evaluated using the Shapiro-Wilk test. For the comparison of the initial and remaining sealer percentages within each group, the Student's t-test was performed. The Kruskal-Wallis test was used to compare the removed sealer percentages among the groups. When a significant difference was detected, pairwise comparisons were performed using the Mann-Whitney U test. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients aged between 18 and 65 years

Patients requiring routine root canal treatment in maxillary first molars

Patients with sufficient cognitive ability to understand and provide informed consent

Teeth undergoing primary root canal treatment

Cases in which the use of an AH Plus epoxy resin-based sealer was deemed appropriate

Exclusion Criteria:

* Teeth with a history of previous root canal treatment

Patients with systemic diseases, known allergies, or pregnancy

Patients who refused to participate or did not provide informed consent

Teeth with unclear visualization of the cavity floor

Cases in which the access cavity design or cleaning protocol could not be standardized

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
preoperative-postoperative macro-photography and photo-based image analysis. | At the time of final access cavity cleaning, immediately following root canal obturation
  For all groups, cleaning effectiveness was measured by comparing pre- and post-cleaning standardized macro photographs of the pulp chamber floor. The percentage of sealer-covered area (SCA) was calculated using pixel-based image analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: ayse karadayi, asst. prof., Principal Investigator — marmara university faculty of dentistry
Locations (1):
- Faculty of Dentistry, Marmara University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided